CLINICAL TRIAL: NCT01166945
Title: Short (5 Days) Versus Long (14 Days) Duration of Antimicrobial Therapy for Acute Bacterial Sinusitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-0452; 130933 (Other: Study Team); H-2010-0129 (Other: HS IRB)
Record Dates: First submitted 2010-07-15; First posted 2010-07-21 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Sinusitis
Keywords: Child; Child, preschool; Sinusitis; Antimicrobial agents
MeSH Terms: conditions — Sinusitis | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short Course (Placebo Comparator): Short course (5 days) of antimicrobial therapy Amoxicillin-Potassium Clavulanate Combination and placebo for next 9 days.
  Interventions: Drug: Amoxicillin-Potassium Clavulanate Combination; Drug: Placebo
- Long Course (Active Comparator): Long course (14 days) of antimicrobial therapy Amoxicillin-Potassium Clavulanate Combination given orally for 14 days.
  Interventions: Drug: Amoxicillin-Potassium Clavulanate Combination

INTERVENTIONS:
Drug: Amoxicillin-Potassium Clavulanate Combination — All subjects will be started on treatment with 5 days of high dose amoxicillin (90mg/kg) with potassium clavulanate (6.4 mg/kg) twice daily in bottle A. The allocation to group B1 or B2 will be concealed until after the family and subject has signed the assent and consent, respectively. The maximum dose will be 2 gms twice daily. After 5 days the subjects will be randomized to either continue to receive the same dose of amoxicillin clavulanate or a look-a-like and taste-a-like placebo for the next 9 days.
  Other Names: there are none
Drug: Placebo — After 5 days the subjects will be randomized to either continue to receive the same dose of amoxicillin clavulanate or a look-a-like and taste-a-like placebo for the next 9 days.
  Other Names: there are none
  Arms: Short Course

SUMMARY:
The investigators objective is to compare short course (5 days) to long course (14 days)antibiotics for the treatment of acute bacterial sinusitis in children. The investigators hypothesize that short course therapy will lead to more frequent relapses of sinusitis and will not reduce resistant organisms.

DETAILED DESCRIPTION:
This was a prospective, randomized, double-blind study comparing short course (5 days) to long course (14 days) antimicrobial therapy for children between 1 and 10 years of age with acute bacterial sinusitis. The major outcome measure is the proportion of children with a clinical relapse on day 10 in the short course therapy group compared to day 20 in the long course therapy group. In addition, the proportion of respiratory flora that are resistant to antibiotics on day 30 will be compared to baseline in each group.

ELIGIBILITY:
Inclusion Criteria:

1. children with nasal discharge (of any quality) or daytime cough (which may be worse at night) or both persisting for 10 days or more without evidence of improvement.
2. families need to be English speaking

Exclusion Criteria:

1. used antibiotics within the last 15 days;
2. had symptoms for > 30 days;
3. have concurrent streptococcal pharyngitis or acute otitis media (as the standard doses for both of these conditions is 10 days);
4. are allergic to penicillin;
5. have symptoms that suggest a complication due to acute bacterial sinusitis that necessitates hospitalization, intravenous antibiotics or sub-specialty evaluation
6. been diagnosed with either immunodeficiency or anatomic abnormality of the upper respiratory tract
7. history of recurrent acute sinusitis (more than 3 episodes in 6 months or 4 episodes in a year)
8. history of chronic sinusitis (more than 90 days of respiratory symptoms in this or the previous respiratory season)
9. girls who have begun menstruating

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2010-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - UW Health Pediatrics (Park St), Madison, Wisconsin
  - UW Health Pediatrics (WestTowne), Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin-Madison Department of Pediatrics Research Information — http://www.pediatrics.wisc.edu/research/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 98 subjects were consented and enrolled. A total of 82 subjects completed the study through day 30. Participants were evaluated on days 5, 10, 15, and 20 for the primary outcome.
Groups:
- Arm A - Short Course Placebo Comparator: Short Course Antibiotic Treatment
  Short course (5 days) of antimicrobial therapy Amoxicillin-Potassium Clavulanate Combination and placebo for next 9 days.
- Arm B - Long Course Treatment: Long Course Antibiotic Treatment
  Long course (14 days) of antimicrobial therapy Amoxicillin-Potassium Clavulanate Combination given orally for 14 days.
Period: Randomized
Arm/Group | Arm A - Short Course Placebo Comparator | Arm B - Long Course Treatment
Started | 51 | 47
Completed | 47 | 43
Not Completed | 4 | 4
Not completed — diagnosed with Group A strep | 4 | 4
Period: Day 5
Arm/Group | Arm A - Short Course Placebo Comparator | Arm B - Long Course Treatment
Started | 47 | 43
Completed | 47 | 43
Not Completed | 0 | 0
Period: Day 10
Arm/Group | Arm A - Short Course Placebo Comparator | Arm B - Long Course Treatment
Started | 47 | 43
Completed | 44 | 41
Not Completed | 3 | 2
Not completed — NonCompliance/Lost to Follow Up | 3 | 2
Period: Day 15
Arm/Group | Arm A - Short Course Placebo Comparator | Arm B - Long Course Treatment
Started | 44 | 41
Completed | 42 | 40
Not Completed | 2 | 1
Not completed — NonCompliance/Lost to Follow Up | 2 | 1
Period: Day 20
Arm/Group | Arm A - Short Course Placebo Comparator | Arm B - Long Course Treatment
Started | 42 | 40
Completed | 42 | 40
Not Completed | 0 | 0
Period: Day 30
Arm/Group | Arm A - Short Course Placebo Comparator | Arm B - Long Course Treatment
Started | 42 | 40
Completed | 38 | 37
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Short Course Antibiotic
- Arm B: Long Course Antibiotic
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 51 | 47 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.7 (2.8) | 5.0 (2.9) | 5.4 (2.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 28 | 23 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 48 | 39 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 22.7 (10.3) | 22.6 (12.2) | 22.65 (11.25)
Temperature at enrollment [Mean (Standard Deviation); unit: celsius] | 110.2 (32.8) | 102.5 (20.6) | 106.4 (26.7)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Children With Clinical Relapse on Day 10 (Short Course) vs Day 20 (Long Course)
Description: Results are based on a daily 6-item symptom survey (day 1 to 14); a daily 3-item survey (day 15 to 30). If a particular symptom is present initially, a score of 2 is given; if it is absent the score is 0. A maximum entry score is 20 (persistent symptoms). If a particular symptom becomes more severe, less severe, or stays the same during treatment, +1, -1, or 0 respectively, will be added to the original score for each symptom. At 10 (and 20 days, respectively), children will be classified as cured, improved or failed based on survey results. Children will be considered cured if they reach a score of < 2. Children will be classified as improved if their score at 10 days (20 days, respectively) is at least 2 points less than their score at 5 days (15 days, respectively). Children will be considered to have failed therapy if their score worsens by + 3 between day 5 (day 15) and day 10 (day 20) or if their score at day 10 (day 20) does not meet criteria for improvement.
Time Frame: at 10 days and at 20 days
Population: 98 participants were enrolled, and 82 completed through day 20. Participant numbers change from day 10 to day 20 due to Group A Strep diagnosis, non-compliance, and lost to follow up over the course of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 51 | 47
Participants
  Day 10: number analyzed (Participants) | 44 | 41
  Day 10: Failed | 13 | 8
  Day 10: Improved | 9 | 10
  Day 10: Cured | 22 | 23
  Day 20: number analyzed (Participants) | 42 | 40
  Day 20: Failed | 16 | 13
  Day 20: Improved | 4 | 3
  Day 20: Cured | 22 | 24

2. Secondary Outcome: Percentage of Participants With Antibiotic Resistant Flora on Day 30 Compared to Baseline
Description: Percentage of participants with antibiotic resistant flora on day 30 compared to baseline
Time Frame: Baseline and 30 days
Population: Number of participants at baseline differed from the number of participants at Day 30 as they were lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Short Course | Long Course
Number analyzed (Participants) | 50 | 46
Participants
  Haemophilis Influenza - Baseline: number analyzed (Participants) | 49 | 46
  Haemophilis Influenza - Baseline | 13 | 13
  Haemophilis Influenza - Day 30: number analyzed (Participants) | 38 | 37
  Haemophilis Influenza - Day 30 | 7 | 5
  Moraxella Catarrhalis - Baseline: number analyzed (Participants) | 49 | 46
  Moraxella Catarrhalis - Baseline | 10 | 13
  Moraxella Catarrhalis - Day 30: number analyzed (Participants) | 38 | 37
  Moraxella Catarrhalis - Day 30 | 11 | 7
  Streptococccus Pneumonia - Baseline: number analyzed (Participants) | 49 | 46
  Streptococccus Pneumonia - Baseline | 11 | 8
  Streptococccus Pneumonia - Day 30: number analyzed (Participants) | 38 | 37
  Streptococccus Pneumonia - Day 30 | 8 | 3
  Streptococcus - Baseline: number analyzed (Participants) | 49 | 46
  Streptococcus - Baseline | 6 | 2
  Streptococcus - Day 30: number analyzed (Participants) | 38 | 37
  Streptococcus - Day 30 | 0 | 0
  Staphylococcus Aureus - Baseline | 2 | 2
  Staphylococcus Aureus - Day 30: number analyzed (Participants) | 38 | 37
  Staphylococcus Aureus - Day 30 | 0 | 1
  No Growth - Baseline: number analyzed (Participants) | 49 | 46
  No Growth - Baseline | 0 | 3
  No Growth - Day 30: number analyzed (Participants) | 38 | 37
  No Growth - Day 30 | 6 | 3
  Other - Baseline: number analyzed (Participants) | 49 | 46
  Other - Baseline | 42 | 36
  Other - Day 30: number analyzed (Participants) | 38 | 37
  Other - Day 30 | 29 | 32

ADVERSE EVENTS:
Time Frame: Days 1 through 30
Groups:
- Arm A: Short Course Antibiotic Treatment
- Arm B: Long Course Antibiotic Treatment
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/47
Other Adverse Events (participants affected / at risk) | 44/51 | 47/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=51) | Arm B (N=47)
Abdominal Pain (Gastrointestinal disorders) | 13 (23) | 21 (30) — Data for number of participants affected is unavailable.
Diarrhea (Gastrointestinal disorders) | 18 (24) | 14 (24) — Data for number of participants affected is unavailable.
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 8 (15) — Data for number of participants affected is unavailable.
Vomiting (Gastrointestinal disorders) | 7 (7) | 13 (17) — Data for number of participants affected is unavailable.

LIMITATIONS AND CAVEATS:
Total number of participants experiencing adverse events is unavailable, the maximum number of participants is reported. The possible range for Arm A is 18-44, the possible range for Arm B is 21-47.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No